CLINICAL TRIAL: NCT06812546
Title: Efficacy and Safety of Early Initiation of Vericiguat in Heart Failure After Acute Myocardial Infarction
Acronym: VIC-MI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dongying Zhang (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other); The First Affiliated Hospital of Chongqing Medical Universty (Unknown)
Responsible Party: Sponsor-Investigator, Dongying Zhang, Professor, Chongqing Emergency Medical Center
Organization: Chongqing Emergency Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIC-MI; 82300372; 82270406 (Other Grant/Funding Number: National Natural Science of Foundation of China); CSTB2024NSCQ-LZX0144 (Other Grant/Funding Number: Chongqing Natural Science Foundation Joint Fund for Innovation and Development); 2022MSXM028 (Other Grant/Funding Number: Chongqing medical scientific research project (Joint project of Chongqing Health Commission and Science and Technolog))
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Acute Myocardial Infarction (AMI); Acute Heart Failure (AHF)
Keywords: Vericiguat; Guideline-Directed Medical Therapy; Heart Failure; Acute myocardial infarction
MeSH Terms: conditions — Heart Failure | interventions — vericiguat

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, prospective, randomized controlled trial in which patients will be randomized into either the experimental or control group by uniform stratification from the main centre.
Who Masked: Outcomes Assessor
Masking Description: The sonographer who interpreted the report, statistician and the investigating physician who completed the 6-minute walk test could not be aware of the grouping of the patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vericiguat Treatment Group (Experimental): Patients enrolled in the experimental group will receive 26 weeks of oral vericiguat on top of the standard treatment, with vericiguat at a dose of 2.5 mg once a day, doubled every fortnight to a maximum dose of 10 mg once a day at the end of week 6 of the visit, which will be maintained for the duration of the treatment.
  Interventions: Drug: Vericiguat
- Standard Treatment Group (No Intervention): Patients enrolled in the controlled group will receive 26 weeks of standard heart failure and coronary heart disease treatment

INTERVENTIONS:
Drug: Vericiguat — Patients enrolled in the experimental group will receive 26 weeks of oral vericiguat on top of the standard treatment, with vericiguat at a dose of 2.5 mg once a day, doubled every fortnight to a maximum dose of 10 mg once a day at the end of week 6 of the visit, which will be maintained for the duration of the treatment.
  Other Names: BAY1021189
  Arms: Vericiguat Treatment Group

SUMMARY:
Heart failure (HF) is a severe cardiovascular disease with extremely high morbidity and mortality rates worldwide, and ischemic cardiomyopathy is an important cause of heart failure. Vericiguat is a soluble guanylate cyclase stimulator which has been verified to improve the cardiovascular outcomes in heart failure patients. The VICTORIA trial excluded patients with acute coronary syndrome in 3 months prior to the study start, so it is still unclear about the efficacy and safety of vericiguat in heart failure after acute myocardial infarction. So we conducted this multi-center, prospective, cohort study to estimate the efficacy and safety of vericiguat in HF patients after acute myocardial infarction.

DETAILED DESCRIPTION:
Heart failure (HF) is a severe cardiovascular disease with extremely high morbidity and mortality rates worldwide, and ischemic cardiomyopathy is an important cause of heart failure. According to different studies, acute heart failure occurs in-hospital in about 14-36% of patients after acute myocardial infarction (AMI)1 and the presence of HF on admission or the occurrence of HF during hospitalization in patients with AMI are strong risk factors for poor prognosis. The incidence of HF in AMI varies according to population differences. For example, in patients with STEMI, the incidence of acute heart failure is relatively high because of the greater extent of the infarction and the longer duration of coronary occlusion, whereas patients with NSTEMI, although at lower risk of developing heart failure in the acute phase, have an increased risk of developing chronic heart failure in the long term. Advanced age, previous history of heart failure, chronic kidney disease, multibranch vasculopathy, and delayed opening of the infarct-related artery are major risk factors. In addition, comorbidities such as diabetes and hypertension increase the risk of developing heart failure.

The goals of treatment for HF after AMI are to improve cardiac function, reduce symptoms, and prevent further myocardial injury. Basic therapy consists of prompt opening of the infarct-related artery (e.g., percutaneous coronary intervention) and the administration of optimized pharmacological treatments such as antiplatelets, beta-blockers, ACEI/ARBs and aldosterone antagonists. In the acute phase, diuretics and positive inotropic agents may be used to relieve severe symptoms. Besides, other HF medication such as SGLT2i are effective in patients with heart failure whether or not it is caused by ischemia.

Vericiguat is a soluble guanylate cyclase stimulator which has been verified to improve the cardiovascular outcomes in heart failure patients. The VICTORIA trial excluded patients with acute coronary syndrome in 3 months prior to the study start, so it is still unclear about the efficacy and safety of vericiguat in heart failure after acute myocardial infarction. The VIC-MI trial is a multi-center, prospective, open-label cohort study to estimate the efficacy and safety of vericiguat in HF patients after acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Undertaking revascularization for criminal coronary artery during hospitalization
* Acute heart failure occurs within 14 days in hospital after STEMI or NSTEMI, meeting all of the following criteria: typical symptoms or signs of heart failure; Treatment with oral or intravenous diuretics is required; LVEF measured by echocardiography is ≤ 45%; Elevated levels of NT proBNP in patients with sinus rhythm ≥ 1000pg/ml and atrial fibrillation/flutter ≥ 1600pg/ml
* eGFR ≥ 15 ml/min/1.73m2
* Informed consent has to be given in written form

Exclusion Criteria:

* Plan to undergo staged revascularization or if the criminal coronary artery has not been successfully opened
* Severe and uncontrolled lung diseases, such as newly developed pulmonary embolism, primary pulmonary hypertension, acute exacerbation of COPD, etc
* Severe liver and kidney dysfunction, Child Pugh grade C or eGFR < 15ml/min/1.73m2
* Allergies to ACEI, ARB, ARNI, beta blockers, SGLT2i, MRA, Vericiguat, and other medications
* Symptomatic hypotension or systolic blood pressure less than 90mmHg after discontinuing intravenous medication
* Women in the perinatal period or those planning to conceive
* Patients planning to undergo elective surgical treatment or tumor chemotherapy
* Diagnosed as Takotsubo cardiomyopathy or nonobstructive acute myocardial infarction (MINOCA)
* Previous diagnosis of cardiomyopathy, including but not limited to dilated cardiomyopathy, hypertrophic cardiomyopathy, etc.
* Autoimmune disease or infectious diseases with typical cardiovascular damage, such as syphilis, systemic lupus erythematosus, etc.
* Diagnosed with severe heart valve disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Serum NT-proBNP Level | Up to 24 weeks
  The primary endpoint of the study is NT-proBNP at the baseline & at the completion of the 24 week intervention

SECONDARY OUTCOMES:
6-minute walk distance | Up to 24 weeks
  6-minute walk distance at the baseline & at the completion of the 24 week intervention
NYHA functional class | Up to 24 weeks
  NYHA functional class at the baseline & at the completion of the 24 week intervention
Worsening heart failure event | Up to 24 weeks
  Time to first worsening heart failure event in 24 weeks after randomization
Left ventricular ejection fraction | Up to 24 weeks
  LVEF measured by echocardiography at the baseline & at the completion of the 24 weeks intervention
Left ventricular end-diastolic diameter | Up to 24 weeks
  LVEDD measured by echocardiography at the baseline & at the completion of the 24 week intervention
Left ventricular global longitudinal strain | Up to 24 weeks
  GLS measured by echocardiography at the baseline & at the completion of the 24 week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, Professor, Study Chair — Chongqing Central Hospital of Chongqing University, Chongqing Emergency Medical Center
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share IPD is not decided yet

REFERENCES:
- [Background] Armstrong PW, Pieske B, Anstrom KJ, Ezekowitz J, Hernandez AF, Butler J, Lam CSP, Ponikowski P, Voors AA, Jia G, McNulty SE, Patel MJ, Roessig L, Koglin J, O'Connor CM; VICTORIA Study Group. Vericiguat in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2020 May 14;382(20):1883-1893. doi: 10.1056/NEJMoa1915928. Epub 2020 Mar 28. PMID 32222134
- [Background] Anker SD, Butler J, Filippatos G, Ferreira JP, Bocchi E, Bohm M, Brunner-La Rocca HP, Choi DJ, Chopra V, Chuquiure-Valenzuela E, Giannetti N, Gomez-Mesa JE, Janssens S, Januzzi JL, Gonzalez-Juanatey JR, Merkely B, Nicholls SJ, Perrone SV, Pina IL, Ponikowski P, Senni M, Sim D, Spinar J, Squire I, Taddei S, Tsutsui H, Verma S, Vinereanu D, Zhang J, Carson P, Lam CSP, Marx N, Zeller C, Sattar N, Jamal W, Schnaidt S, Schnee JM, Brueckmann M, Pocock SJ, Zannad F, Packer M; EMPEROR-Preserved Trial Investigators. Empagliflozin in Heart Failure with a Preserved Ejection Fraction. N Engl J Med. 2021 Oct 14;385(16):1451-1461. doi: 10.1056/NEJMoa2107038. Epub 2021 Aug 27. PMID 34449189
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Juilliere Y, Cambou JP, Bataille V, Mulak G, Galinier M, Gibelin P, Benamer H, Bouvaist H, Meneveau N, Tabone X, Simon T, Danchin N; FAST-MI Investigators. Heart failure in acute myocardial infarction: a comparison between patients with or without heart failure criteria from the FAST-MI registry. Rev Esp Cardiol (Engl Ed). 2012 Apr;65(4):326-33. doi: 10.1016/j.recesp.2011.10.027. Epub 2012 Feb 20. PMID 22357361
- [Background] Bahit MC, Lopes RD, Clare RM, Newby LK, Pieper KS, Van de Werf F, Armstrong PW, Mahaffey KW, Harrington RA, Diaz R, Ohman EM, White HD, James S, Granger CB. Heart failure complicating non-ST-segment elevation acute coronary syndrome: timing, predictors, and clinical outcomes. JACC Heart Fail. 2013 Jun;1(3):223-9. doi: 10.1016/j.jchf.2013.02.007. Epub 2013 Jun 3. PMID 24621874
- [Background] Steg PG, Dabbous OH, Feldman LJ, Cohen-Solal A, Aumont MC, Lopez-Sendon J, Budaj A, Goldberg RJ, Klein W, Anderson FA Jr; Global Registry of Acute Coronary Events Investigators. Determinants and prognostic impact of heart failure complicating acute coronary syndromes: observations from the Global Registry of Acute Coronary Events (GRACE). Circulation. 2004 Feb 3;109(4):494-9. doi: 10.1161/01.CIR.0000109691.16944.DA. Epub 2004 Jan 26. PMID 14744970
- [Background] Bahit MC, Kochar A, Granger CB. Post-Myocardial Infarction Heart Failure. JACC Heart Fail. 2018 Mar;6(3):179-186. doi: 10.1016/j.jchf.2017.09.015. PMID 29496021